CLINICAL TRIAL: NCT05032027
Title: A Randomized Controlled Clinical Study of Oral Probiotics on Radiation Enteritis Stage Ⅱ Induced by Pelvic Concurrent Chemoradiotherapy
Brief Title: Oral Probiotics on Radiation Enteritis Stage Ⅱ Induced by Pelvic Concurrent Chemoradiotherapy
Acronym: probiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JCL2021-1
Record Dates: First submitted 2021-06-23; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-06

CONDITIONS: Pelvic Cancer, Enteritis, Probiotics,Chemoradiotherapy
MeSH Terms: conditions — Pelvic Neoplasms; Enteritis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The random assignment of patients was performed by Nanchang Medical University with a computer-generated random number code. Patients were randomly distributed in a 1:1 ratio to receive probiotics or a placebo (the block size was known only to the statistician). The drug was distributed and packaged in accordance with random numbers, and the documents stating the parameters, such as the blinding codes for the seeds of the random numbers, the block length, and the random numbers, were sealed in envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic group (Experimental): Probiotic( recieving Probiotic at the first day of chemoradiotherapy daily)with radiotherapy and Chemotherapy Intervention
  Interventions: Other: probiotics
- placebo group (No Intervention): placebo( one times a day)with radiotherapy and Chemotherapy Intervention
- healthy control group (No Intervention): healthy control group

INTERVENTIONS:
Other: probiotics — recieving probiotics at the first day of chemoradiotherapy daily
  Arms: Probiotic group

SUMMARY:
Effect of Probiotics on Raditon Enteritis in Pelvic Tumor Patients Receiving Radiotherapy.

DETAILED DESCRIPTION:
Radiation-induced enteritis is an common and severe side effect of the patients undergoing pelvic radiotherapy. It can lead to dose-limiting and debilitating treatment effect. There is no guideline on an acknowledged intervention that significantly reduces its severity. In previous study, we have abserved that a probiotic combination significantly enhances the immune response of patients and reduces the severity of oral mucositis through modification of gut microbiota. In this stuyd we plan to designe a randomized trial of Probiotics probiotics in patients with pelvic carcinoma.The aim of this study is to determine if regulating intestinal tract flora will reduce the severity of radiation-induced mucositis in patients receiving pelvic radiotherapy. The effect of this intervention on a patient's general well-being was also investigated. The primary end-point of the study was the incidence of grade 3 enteritis. In 2021, 40 patients are estimated to be recruited into the study in Jiangxi Cancer Hospitals, China. 20 patients were randomized to receive Probiotics or placebo during chemoradiotherapy respectively.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky score ≥80 pelvic tumor patients receiving chemoradiotherapy in our Cancer Center

Exclusion Criteria:

* any immune system disease under high risk to antimicrobial agents such as Diabetes,infection disease or drug allergy to Probiotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-27 (Estimated); Primary Completion 2022-12-27 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
grade 3 entiritis | one month
  Diarrhea more than seven times a day

SECONDARY OUTCOMES:
AE | one month
  Adverse drug events
immune index | one month
  immune globulin
Changes in intestinal flora | one month
  Dung sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, MD,PHD, Principal Investigator — radiation department of Jiangxi cancer hospital
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided